CLINICAL TRIAL: NCT01103960
Title: 8 Week Randomised Double-blind Study to Compare the Efficacy and Safety of Telmisartan 80mg+ Amlodipine 5 mg vs. Amlodipine 5mg Monotherapy in Patients With Hypertension Who Fail to Respond Adequately to Treatment With Amlodipine 5mg Monotherapy
Brief Title: An Eight-week Randomized,Double-blind Study to Evaluate the Efficacy and Safety of Fixed-dose Combinations of T80+A5 Versus A5 Monotherapy in Patients With Hypertension Who Fail to Respond Adequately to Treatment With A5 Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1235.29
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

ARMS (2):
- Telmisartan80mg+Amlodipine5mg (Experimental): combination therapy
  Interventions: Drug: Telmisartan80mg+Amlodipine5mg
- amlodipine 5 mg (Active Comparator): Monotherapy
  Interventions: Drug: amlodipine 5mg; Drug: Telmisartan80mg+Amlodipine 5mg

INTERVENTIONS:
Drug: Telmisartan80mg+Amlodipine5mg — combination therapy
  Arms: Telmisartan80mg+Amlodipine5mg
Drug: amlodipine 5mg — monotherapy
  Arms: amlodipine 5 mg
Drug: Telmisartan80mg+Amlodipine 5mg — combination therapy
  Arms: amlodipine 5 mg

SUMMARY:
The primary objectives of this trial is to demonstrate that the fixed-dose combination of telmisartan 80mg plus amlodipine 5mg (T80/A5) is superior to amlodipine 5mg (A5) in reducing seated trough diastolic blood pressure (DBP) at 8 weeks.

ELIGIBILITY:
Inclusion criteria:

1. diagnosis of essential hypertension
2. failure to respond adequately to six weeks treatment with amlodipine 5 mg monotherapy
3. provision of written informed consent

Exclusion criteria:

1. clinical conditions which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of telmisartan and amlodipine for the planned duration of this trial (e.g. populations where labeling of either product recommends against its utilization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- China (12):
  - 1235.29.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1235.29.86004 Boehringer Ingelheim Investigational Site, Beijing
  - 1235.29.86006 Boehringer Ingelheim Investigational Site, Changchun
  - 1235.29.86013 Boehringer Ingelheim Investigational Site, Changsha
  - 1235.29.86014 Boehringer Ingelheim Investigational Site, Guangzhou
  - 1235.29.86012 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1235.29.86002 Boehringer Ingelheim Investigational Site, Shanghai
  - 1235.29.86009 Boehringer Ingelheim Investigational Site, Shanghai
  - 1235.29.86010 Boehringer Ingelheim Investigational Site, Shanghai
  - 1235.29.86011 Boehringer Ingelheim Investigational Site, Shanghai
  - 1235.29.86007 Boehringer Ingelheim Investigational Site, Shenyang
  - 1235.29.86008 Boehringer Ingelheim Investigational Site, Tianjin
- Malaysia (2):
  - 1235.29.60017 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 1235.29.60016 Boehringer Ingelheim Investigational Site, Kuala Lumpur
- Philippines (2):
  - 1235.29.63018 Boehringer Ingelheim Investigational Site, Metro Manila
  - 1235.29.63019 Boehringer Ingelheim Investigational Site, Quezon City

REFERENCES:
- [Derived] Zhu D, Gao P, Holtbruegge W, Huang C. A randomized, double-blind study to evaluate the efficacy and safety of a single-pill combination of telmisartan 80 mg/amlodipine 5 mg versus amlodipine 5 mg in hypertensive Asian patients. J Int Med Res. 2014 Feb;42(1):52-66. doi: 10.1177/0300060513503756. Epub 2014 Jan 3. PMID 24391142

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Whilst there were 324 patients randomised and treated, there were only 314 in the Full analysis set (FAS).
Groups:
- A5 Alone: Amlodipine 5mg monotherapy
- T80/A5: Telmisartan 80mg plus Amlodipine 5mg fixed-dose combination
Period: Overall Study
Arm/Group | A5 Alone | T80/A5
Started | 164 (Randomised and treated.) | 160 (Randomised and treated.)
Completed | 159 (Completed study medication.) | 158 (Completed study medication.)
Not Completed | 5 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A5 Alone | T80/A5 | Total
Number analyzed (Participants) | 159 | 155 | 314
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (9.7) | 52.4 (8.7) | 52.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 78 | 149
  Male | 88 | 77 | 165
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 97.84 (6.43) | 97.21 (5.46) | 97.53 (5.97)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 146.27 (11.15) | 146.44 (12.20) | 146.35 (11.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DBP After 8 Weeks of Treatment
Description: Seated trough DBP after 8 weeks or last observation carried forward (LOCF). Analysis will be adjusted for treatment, country, and baseline measurement of endpoint.
Time Frame: Baseline and 8 weeks
Population: Full analysis set (FAS) defined as patients randomised, treated, with a baseline endpoint measurement and at least one post-dose endpoint measurement during the double blind (DB) phase.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 159 | 155
mmHg | -10.19 (0.93) | -12.38 (0.95)
Statistical Analysis 1: Comparison: A5 Alone vs T80/A5; A5 minus T80/A5; Test type: Superiority or Other; p = 0.007, ANCOVA — This was the first step in the closed testing procedure of multiple endpoints. The p-value was <0.05 so this test was considered confirmatory. Proceeding to the next step was allowed, testing the same endpoint in the subgroup of Chinese patients; Mean Difference (Final Values) = 2.1881, 95% CI [0.6082 to 3.7681], Standard Error of Mean 0.8030

2. Primary Outcome: Change From Baseline in DBP After 8 Weeks of Treatment in Chinese Patients
Description: Seated trough DBP after 8 weeks or LOCF in Chinese patients. Analysis will be adjusted for treatment and baseline measurement of endpoint.
Time Frame: Baseline and 8 weeks
Population: FAS with LOCF and further restricted to the Chinese subgroup
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 133 | 129
mmHg | -8.85 (0.63) | -10.77 (0.64)
Statistical Analysis 1: Comparison: A5 Alone vs T80/A5; A5 minus T80/A5; Test type: Superiority or Other; p = 0.034, ANCOVA — This was the second step in the closed testing procedure of multiple endpoints. The p-value was again <0.05 so this test was also considered confirmatory; Mean Difference (Final Values) = 1.9195, 95% CI [0.1443 to 3.6947], Standard Error of Mean 0.9015

3. Secondary Outcome: Change From Baseline in SBP After 8 Weeks of Treatment
Description: Seated trough SBP after 8 weeks or LOCF. Analysis will be adjusted for treatment, country, and baseline measurement of endpoint.
Time Frame: Baseline and 8 weeks
Population: FAS with LOCF
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 159 | 155
mmHg | -11.66 (1.30) | -16.15 (1.33)
Statistical Analysis 1: Comparison: A5 Alone vs T80/A5; A5 minus T80/A5; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.4879, 95% CI [2.2807 to 6.6950], Standard Error of Mean 1.1217

4. Secondary Outcome: DBP and SBP Control and Response After 8 Weeks of Treatment
Description: DBP control is defined as DBP <90 mmHg or <80 mmHg in patients with diabetes or renal impairment. SBP control is defined as SBP <140 mmHg or <130 mmHg in patients with diabetes or renal impairment. DBP response is defined as DBP <90 mmHg or <80 mmHg in patients with diabetes or renal impairment or a reduction from baseline >=10mmHg. SBP response is defined as SBP<140 mmHg or <130 mmHg in patients with diabetes or renal impairment or a reduction from baseline >=15mmHg.
Time Frame: Baseline and 8 weeks
Population: FAS with LOCF
Measure: Number; unit: Number of participants
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 159 | 155
Number of participants
  DBP control | 85 | 112
  SBP control | 100 | 119
  DBP response | 101 | 124
  SBP response | 120 | 131

5. Secondary Outcome: Number of Patients in Blood Pressure Categories Over Time
Description: BP optimal: SBP <120 mmHg and DBP <80 mmHg, BP normal: SBP <130 mmHg and DBP <85 mmHg but not optimal, BP high-normal: SBP <140 mmHg and DBP <90 mmHg but not normal. Grade 1 hypertension: SBP <160 mmHg and DBP <100 mmHg but not high-normal, Grade 2 hypertension: SBP <180 mmHg and DBP <110 mmHg but not grade 1, Grade 3 hypertension: SBP >=180 mmHg or DBP >=110 mmHg.
Time Frame: 8 weeks
Population: FAS with LOCF
Measure: Number; unit: Number of participants
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 159 | 155
Number of participants
  BP optimal | 7 | 11
  BP normal | 33 | 36
  BP high-normal | 32 | 53
  Grade 1 hypertension | 69 | 48
  Grade 2 hypertension | 15 | 5
  Grade 3 hypertension | 3 | 2

6. Secondary Outcome: Change From Baseline in DBP After 4 Weeks of Treatment
Description: Seated trough DBP after 4 weeks.
Time Frame: Baseline and 4 weeks
Population: FAS with LOCF
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 158 | 155
mmHg | -7.51 (6.80) | -9.41 (7.26)

7. Secondary Outcome: Change From Baseline in SBP After 4 Weeks of Treatment
Description: Seated trough SBP after 4 weeks.
Time Frame: Baseline and 4 weeks
Population: FAS with LOCF
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 158 | 155
mmHg | -8.19 (11.45) | -12.10 (11.68)

8. Secondary Outcome: DBP and SBP Control and Response After 4 Weeks of Treatment
Description: as for outcome 4
Time Frame: Baseline and 4 weeks
Population: FAS with LOCF
Measure: Number; unit: Number of participants
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 159 | 155
Number of participants
  DBP control | 71 | 95
  SBP control | 91 | 103
  DBP response | 87 | 108
  SBP response | 108 | 124

9. Secondary Outcome: Number of Patients in Blood Pressure Categories at 4 Weeks
Description: as for outcome 5
Time Frame: 4 weeks
Population: FAS with LOCF
Measure: Number; unit: Number of participants
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 159 | 155
Number of participants
  BP optimal | 1 | 7
  BP normal | 20 | 26
  BP high-normal | 35 | 44
  Grade 1 hypertension | 81 | 62
  Grade 2 hypertension | 17 | 15
  Grade 3 hypertension | 5 | 1

10. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Pulse Rate, Laboratory Parameters and ECG.
Description: Clinically relevant abnormalities for Physical examination, pulse rate, laboratory parameters and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: From drug administration until end of treatment plus one day
Population: Treated set included patients who were randomised and took at least one dose of the trial medication in the double-blind treatment period.
Measure: Number; unit: participants
Arm/Group | A5 Alone | T80/A5
Number analyzed (Participants) | 164 | 160
participants
  Atrial fibrilation | 0 | 1
  Myocardial ischaemia | 1 | 0
  Blood glucose increased | 1 | 4
  Protein urine present | 2 | 1
  Alanine aminotransferase increased | 0 | 1
  Blood creatinine phosphokinase increased | 1 | 0
  Blood creatinine increased | 0 | 1
  Blood glucose abnormal | 1 | 1
  Heart rate increased | 0 | 1

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- A5 Alone: Amlodipine 5 mg one daily
- T80/A5: Telmisartan 80 mg plus Amlodipine 5 mg once daily
Arm/Group | A5 Alone | T80/A5
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/160
Other Adverse Events (participants affected / at risk) | 0/164 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.